CLINICAL TRIAL: NCT04872257
Title: Combined Therapy With NB-UVB Phototherapy and Oral Vitamin D Supplementation in Patients With Vitiligo: a Randomized-clinical Trial, Triple-blind, Placebo-controlled
Brief Title: Oral Vitamin D Supplementation Combined With Phototherapy as a Treatment for Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Jorge Valdespino Valdes, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DE19-00002
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Vitiligo; Vitiligo, Generalized; Autoimmune; Autoimmune Diseases; Autoimmune Disease Skin
Keywords: vitiligo; randomized clinical trial; vitamin D; phototherapy; quality of life
MeSH Terms: conditions — Vitiligo; Autoimmune Diseases | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Our randomization and blinding process is in charge by a nurse who is not part of the study. A pharmacy school laboratory (not part of the study) randomly assigned the intervention and placebo to each patient (1-20) as treatment A or B. This information was delivered in a sealed envelope, in which only the nurse had access to. Neither the participants, investigators and outcome assessor, nor the data analyst know which patient is receiving the experimental treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Vitamin D + NB-UVB Phototherapy (Experimental)
  Interventions: Drug: Oral Vitamin D; Procedure: NB-UVB Phototherapy
- Placebo + NB-UVB Phototherapy (Placebo Comparator)
  Interventions: Procedure: NB-UVB Phototherapy; Drug: Placebo

INTERVENTIONS:
Drug: Oral Vitamin D — Vitamin D 5,000 UI for 6 months (oral capsule, daily, single-dose)
  Arms: Oral Vitamin D + NB-UVB Phototherapy
Procedure: NB-UVB Phototherapy — NB-UVB Phototherapy twice per week for 6 months until completing 48 sessions. Initial dose of 200 mJ/cm² with a 10-20% increase to the previous session. Maximum dose for face and neck is 1500 mJ/cm² and 3000 mJ/cm² for the rest of the body.
Drug: Placebo — Administered orally daily for 6 months
  Arms: Placebo + NB-UVB Phototherapy

SUMMARY:
A randomized clinical trial that treats vitiligo patients with oral vitamin D and Narrow-Band Ultraviolet B (NB-UVB) phototherapy (intervention group); or placebo and NB-UVB phototherapy (control group). We will evaluate if the group supplemented with vitamin D achieves a higher repigmentation rate than the control group, proving the relevance of vitamin D as an immunomodulator in the pathophysiology of vitiligo. These findings may support the use of vitamin D as an economic, safe, and adjuvant treatment for vitiligo.

DETAILED DESCRIPTION:
A randomized clinical trial, triple-blind, placebo-controlled treating patients with diagnosed vitiligo. The intervention group will be treated with oral vitamin D 5,000 IU per day and NB-UVB phototherapy. The control group will be treated with placebo and NB-UVB phototherapy. We will evaluate the efficacy (repigmentation rate) and improvement of the quality of life with vitamin D and phototherapy versus placebo and phototherapy.

Our objectives are:

* Evaluate if the use of the supplementation with oral vitamin D accelerates the repigmentation rate in vitiligo lesions treated with NB-UVB phototherapy, achieving a lower accumulated dose of phototherapy.
* Compare basal blood levels of vitamin D before and after treatment completion.
* Compare quality of life of the intervention group with the control group.
* Associate pigmentation rates between intervention and control group obtained with tools that assess activity of disease, such as, Vitiligo Area and Severity Index (VASI) and Vitiligo European Task Force (VETF) score.
* Compare results in quality of life between intervention and control group obtained with tools, such as, Vitiligo-Specific Quality-of-Life Instrument (VitiQoL) and Dermatology Life Quality Index (DLQI).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age at the time of signing the informed consent document.
* ≥5% of affected skin area
* Inactive, generalized vitiligo (inactive for a minimum of 6 months). [Inactive: No new spontaneous lesions or a rapid progression of these.]
* Subjects who have not been treated with phototherapy previously.
* Subject who have not been treated with topical corticosteroids for at least 8 weeks or immunomodulators for at least 12 weeks.

Exclusion Criteria:

* Subjects with <5% of affected skin area
* Subjects who use multivitamins, diuretics, lipase-inhibitors (orlistat)
* Subjects with calcium disorders (for example: primary hyperparathyroidism) or patients with hepatic/kidney failure.
* Subjects with malabsorption gastrointestinal disorders
* Pregnant women or in lactation
* Subjects with cancer
* Subjects with previous history of skin cancer (melanoma/non-melanoma)
* Photo-sensible diseases (actinic dermatitis, porphyria, xeroderma pigmentosa) or drugs
* Subjects using immunomodulator o immunosuppressor treatments
* Subjects who practice activities that require prolonged sun exposure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
VASI score - Vitiligo Area and Severity Index (VASI) | Week 0
  The VASI score is used to assess the severity and extent of Vitiligo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
VASI score - Vitiligo Area and Severity Index (VASI) | Week 12
  The VASI score is used to assess the severity and extent of Vitiligo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
VASI score - Vitiligo Area and Severity Index (VASI) | Week 24
  The VASI score is used to assess the severity and extent of Vitiligo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.

SECONDARY OUTCOMES:
VETF score - Vitiligo European Task Force (VETF) score | Week 0
  The VETF is a validated scoring system that assesses 3 dimensions of the disease (extent, staging, and spreading/progression). (1) the extent of vitiligo will be estimated as the percentage of vitiligo involvement of 5 body sites. (2) Stage of vitiligo will be assessed as 0 (normal pigmentation), 1 (incomplete depigmentation), 2 (complete depigmentation), 3 (partial hair whitening [<30%]), and 4 (complete hair whitening). (3) Spreading of vitiligo will be scored as 0 (stable disease), -1 (observed ongoing subclinical repigmentation), and +1 (additional patches in a given area or observed ongoing subclinical depigmentation). The VETF score calculated as follows:
  VETF Extent or Staging or Spreading = Sum of all specific values for that category from all body sites (% of Area affected for Extent; 0-20 for Staging; -5 to +5 for Spreading).
VETF score - Vitiligo European Task Force (VETF) score | Week 12
  The VETF is a validated scoring system that assesses 3 dimensions of the disease (extent, staging, and spreading/progression). (1) the extent of vitiligo will be estimated as the percentage of vitiligo involvement of 5 body sites. (2) Stage of vitiligo will be assessed as 0 (normal pigmentation), 1 (incomplete depigmentation), 2 (complete depigmentation), 3 (partial hair whitening [<30%]), and 4 (complete hair whitening). (3) Spreading of vitiligo will be scored as 0 (stable disease), -1 (observed ongoing subclinical repigmentation), and +1 (additional patches in a given area or observed ongoing subclinical depigmentation). The VETF score calculated as follows:
  VETF Extent or Staging or Spreading = Sum of all specific values for that category from all body sites (% of Area affected for Extent; 0-20 for Staging; -5 to +5 for Spreading).
VETF score - Vitiligo European Task Force (VETF) score | Week 24
  The VETF is a validated scoring system that assesses 3 dimensions of the disease (extent, staging, and spreading/progression). (1) the extent of vitiligo will be estimated as the percentage of vitiligo involvement of 5 body sites. (2) Stage of vitiligo will be assessed as 0 (normal pigmentation), 1 (incomplete depigmentation), 2 (complete depigmentation), 3 (partial hair whitening [<30%]), and 4 (complete hair whitening). (3) Spreading of vitiligo will be scored as 0 (stable disease), -1 (observed ongoing subclinical repigmentation), and +1 (additional patches in a given area or observed ongoing subclinical depigmentation). The VETF score calculated as follows:
  VETF Extent or Staging or Spreading = Sum of all specific values for that category from all body sites (% of Area affected for Extent; 0-20 for Staging; -5 to +5 for Spreading).
Vitamin D blood levels | Week 0
  Measure vitamin D levels on blood between the intervention and control group
Vitamin D blood levels | Week 12
  Measure vitamin D levels on blood between the intervention and control group
Vitamin D blood levels | Week 24
  Measure vitamin D levels on blood between the intervention and control group
DLQI - Dermatology Life Quality Index | Week 0
  The DLQI is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions, and its use has been described in over 1000 publications including many multinational studies. The DLQI is the most frequently used instrument in studies of randomized controlled trials in dermatology.
DLQI - Dermatology Life Quality Index | Week 24
  The DLQI is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions, and its use has been described in over 1000 publications including many multinational studies. The DLQI is the most frequently used instrument in studies of randomized controlled trials in dermatology.
VitiQoL - Vitiligo Specific Quality of Life | Week 0
  VitiQoL is an instrument specific for vitiligo that consists of 16 items, in which the patient perceives the severity of their disease and how it affects their quality of life.
VitiQoL - Vitiligo Specific Quality of Life | Week 24
  VitiQoL is an instrument specific for vitiligo that consists of 16 items, in which the patient perceives the severity of their disease and how it affects their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian B Cuellar-Barboza, MD, Principal Investigator — Hospital Universitario "Dr. Jose Eleuterio Gonzalez"
Locations (1):
- Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No